CLINICAL TRIAL: NCT05817942
Title: A Prospective, Non-interventional, Multi-country Cohort Study of the Effectiveness and Safety of Filgotinib in Adult Patients With Moderately to Severely Active Ulcerative Colitis
Brief Title: Prospective Observational Study of Effectiveness and Safety of Filgotinib in Participants With Ulcerative Colitis (UC)
Acronym: GALOCEAN
Status: Active, not recruiting | Type: Observational
Sponsor: Alfasigma S.p.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: GLPG0634-CL-425; 105477 (Other: HMA-EMA Catalogues)
Record Dates: First submitted 2023-04-05; First posted 2023-04-18 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Ulcerative Colitis
Keywords: filgotinib; safety; efficacy
MeSH Terms: conditions — Colitis, Ulcerative | interventions — GLPG0634

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Arm A: Filgotinib: Participants diagnosed with moderately or severely active UC taking filgotinib according to local treatment guidelines or routine clinical practice and product information.
  Interventions: Drug: Filgotinib

INTERVENTIONS:
Drug: Filgotinib — Jyseleca

SUMMARY:
To describe the effectiveness, treatment patterns, quality of life, and safety of participants with moderately or severely active UC treated with filgotinib in a real-world setting.

ELIGIBILITY:
Inclusion Criteria:

1. Filgotinib-naïve participants with moderately or severely active UC as judged by the physician and starting filgotinib treatment according to local treatment guidelines, routine practices and product information.

Exclusion Criteria:

1. Participation in any interventional or non-interventional study without prior approval from the medical leader. This does not preclude inclusion of participants enrolled to national registries.
2. Participant is diagnosed with Crohn's disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of participants aged 18 years or older with moderately or severely active UC as judged by the physician and starting filgotinib treatment. Participants are enrolled across around 10 countries in Europe, including the United Kingdom.
Sampling Method: Non-Probability Sample
Enrollment: 509 (Actual)
Dates: Start 2023-06-12 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Treatment Persistence Rate at week 52. | Week 52
  The persistence rate is defined as the percentage of participants who have continued filgotinib treatment since initiation.

SECONDARY OUTCOMES:
Treatment Persistence Rate at weeks 10, 24, 76 and 104 | Weeks 10, 24, 76 and 104
Clinical Response Rate | Weeks 10, 24, 52, 76 and 104
Clinical Remission Rate | Weeks 10, 24, 52, 76 and 104
Change from Baseline in Health-Related Quality of Life (HRQoL) as measured by the Short Inflammatory Bowel Disease Questionnaire (SIBDQ) | Baseline, Weeks 10, 24, 52, 76 and 104
Change from Baseline in HRQoL as measured by the Urgency Numeric Rating Scale (NRS) | Baseline, Weeks 10, 24, 52
Change from Baseline in HRQoL as measured by the Functional Assessment of Chronic Illness Therapy-Fatigue score (FACIT-F) | Baseline, Weeks 10, 24, 52, 76 and 104
Number of Participants with Adverse Events (AEs) | Up to 104 Weeks
Number of Participants with Serious Adverse Events (SAEs) | Up To 104 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Alfasigma Study Director, Study Director — Alfasigma S.p.A.
Locations (81):
- Austria (4):
  - LKH - Universitätsklinikum Graz, Graz
  - Klinikum Klagenfurt am Wörthersee, Klagenfurt
  - KH der Barmherzigen Brüder St.Veit an der Glan, Sankt Veit an der Glan
  - AKH - Medizinische Universität Wien, Vienna
- Belgium (12):
  - Imeldaziekenhuis, Bonheiden
  - CHU Saint-Pierre, Brussels
  - Cliniques Universitaires de Bruxelles Hopital Erasme, Brussels
  - UZA, Edegem
  - AZ Maria Middelares, Ghent
  - AZ Sint-Lucas, Ghent
  - Universitair Ziekenhuis Gent, Ghent
  - Sint-Franciscus ziekenhuis, Heusden-Zolder
  - UZ Leuven, Leuven
  - CHU de Liège, Liège
  - Clinique CHC MontLégia, Liège
  - AZ Damiaan, Ostend
- France (13):
  - CHU Amiens - Hopital Sud, Amiens
  - Hôpital Jean Minjoz, Besançon
  - Clinique Abroise Paré, Clichy
  - CHU de Grenoble - Hôpital Nord, Grenoble
  - CHU Lille - Hôpital Claude Huriez, Lille
  - CHU Montpellier- Hôpital Saint Eloi, Montpellier
  - CHRU de Nancy, Nancy
  - CHU Nantes - Hôtel Dieu, Nantes
  - Hôpital Saint-Louis, Paris
  - CHU Bordeaux - Hôpital Haut-Lévêque, Pessac
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHU Saint Etienne - Hôpital Nord, Saint-Etienne
  - Hôpital Rangueil, Toulouse
- Germany (10):
  - Synesis GmbH, Grünwald, Bavaria
  - Klinikum St. Marien Amberg, Amberg
  - Medizinisches Versorgungszentrum Dachau, Dachau
  - Fachinternistische Schwerpunktpraxis, Hamburg
  - Praxis fur Gastroenterologie, Heidelberg
  - Universitaetsklinikum Schleswig-Holstein, Kiel
  - Universitätsklinikum Leipzig AöR, Leipzig
  - Gastro Campus Research GbR, Münster
  - Magen-Darm-Zentrum Remscheid, Remscheid
  - Universitätsklinikum Tübingen, Tübingen
- Ireland (3):
  - Cork University Hospital, Cork
  - St Vincent's University Hospital, Dublin
  - Beaumont Hospital, Dublin
- Italy (9):
  - Azienda Ospedaliera Saverio De Bellis - Castellana Grotte, Bari, Italia
  - IRCCS Ospedale San Raffaele ,Via Olgettina 60, Milan, Italia
  - Azienda Ospedaliero Universitaria Pisana - Cisanello, Pisa, Italia
  - Fondazione IRCCS CA' Granda Ospedale Maggiore Policlinico, Milan
  - ASST Fatebenefratelli Sacco, Milan
  - IRCCS Ospedale Sacro Cuore Don Calabria, Negrar
  - Azienda Ospedaliera Ospedali Riuniti Villa Sofia - Cervello, Palermo
  - IRCCS Istituto Clinico Humanitas, Rozzano
  - Ospedale Mauriziano Umberto I, Torino
- Netherlands (8):
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Amsterdam UMC (AMC), Amsterdam
  - Zuyderland Medisch Centrum - Sittard-Geleen, Geleen
  - Radboud UMC, Nijmegen
  - Erasmus MC, Rotterdam
  - Franciscus Gasthuis, Rotterdam
  - ETZ Elisabeth, Tilburg
  - UMC Utrecht, Utrecht
- Norway (6):
  - Nordlandsykehuset, Bodø
  - Akershus Universitetssykehus, Lørenskog
  - Oslo University Hospital, Oslo
  - Bærum Hospital , Gjettum, Oslo
  - Universitetssykehuset Nord-Norge, Tromsø
  - St. Olav's University Hospital, Trondheim
- Spain (6):
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Catalonia
  - Hospital Universitari Germans Trias i Pujol, Badalona, Spain
  - Hospital Clinic de Barcelona, C/ Villarroel, 170, Barcelona, Spain
  - Hospital Universitario de Gran Canaria Dr. Negrin, Las Palmas de Gran Canaria, Spain
  - Hospital Universitari Son Espases, Palma de Mallorca, Spain
  - Hospital Universitario de Santiago de Compostela, Santiago de Compostela, Spain
- United Kingdom (10):
  - The Ulster Hospital, Belfast
  - Bury Care Organisation, Bury
  - Royal Devon University Healthcare NHS Foundation trust, Exeter
  - Glasgow Royal Infirmary, Glasgow
  - Queen Elizabeth University Hospital, Glasgow
  - St Mark's Hospital, Central Middlesex, Acton Lane, London
  - St George's Hospital, London
  - Norfolk and Norwich University Hospital, Norwich
  - John Radcliffe Hospital, Oxford
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: No